CLINICAL TRIAL: NCT06315959
Title: Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Chronic Pain Following Open Heart Surgery: A Prospective Randomized Controlled Trial
Brief Title: Bilateral Erector Spinae Plane Block for Postoperative Chronic Pain After Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESPCHRONIC2023
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain; Cardiac Surgery; Post Operative Pain
Keywords: Chronic Pain; Cardiac surgery; Erector Spinae Plane Block
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative | interventions — Passive Cutaneous Anaphylaxis; Control Groups

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program, 'Research Randomizer (Urbaniak and Plous, 2013)'.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes containing study participation numbers will be used to assign each patient. A researcher not involved in patient follow-up will use the web-based "Research Randomizer" (Urbaniak and Plous 2013) tool to give each participation number to a random group with a 1:1 ratio. A nurse not an active investigator in the study will have each participant choose an envelope containing the study participation number. They will inform the anesthetist administering the block/blocks about which group the patient is in immediately before administration. Researchers, surgeons, and nurses will not be aware of the randomization of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESP (Active Comparator): A bilateral ESP Block(60 ml, %0.25 bupivacaine, totally) + IV morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: Bilateral ultrasound guided erector spinae plane block; Drug: morphine PCA
- Group Control (Other): IV morphine PCA
  Interventions: Other: Control group; Drug: morphine PCA

INTERVENTIONS:
Procedure: Bilateral ultrasound guided erector spinae plane block — Bilateral ultrasound-guided ESP(total of 60 ml, %0.25 bupivacaine) will be performed + IV morphine PCA Multimodal analgesia : Intraoperatively, all patients will receive 0.05 mg/kg (IBW) iv morphine. Thirty minutes before the end of surgery, 1 gram of intravenous paracetamol will be administered. Postoperative analgesia: iv paracetamol 1gr every 8 hours and IV PCA of 0,5mg/ml morphine. In cases where rescue analgesia is required (NRS score ≥4),iv fentanyl 25-50 mcg and/or ibuprofen and/or ketamine 10 mg will be administered. Patients are routinely administered iv dexamethasone 4 mg and IV 8 mg ondansetron 20 minutes before end of surgery for postoperative nausea and vomiting prophylaxis.
  Postoperative chronic pain will be assessed using the Brief Pain Inventory(BPI).
  Anxiety and depression status will be evaluated using the Hospital Anxiety and Depression Scale (HADS).
  The character of pain will be evaluated using the Douleur Neuropathique 4 (DN4) score.
  Other Names: erector spinae plane block
  Arms: Group ESP
Drug: morphine PCA — IV PCA of 0,5mg/ml morphine (the bolus dose is 20 µg/kg, the lock-in time of 6-10 minutes, the 4-hour limit is adjusted to be 80% of the calculated total amount).
  Other Names: PCA
  Arms: Group ESP
Other: Control group — Patients in this group will not be performed plane blocks. Multimodal analgesia : Intraoperatively, all patients will receive 0.05 mg/kg (IBW) iv morphine. Thirty minutes before the end of surgery, 1 gram of intravenous paracetamol will be administered. Postoperative analgesia: iv paracetamol 1gr every 8 hours and IV PCA of 0,5mg/ml morphine. In cases where rescue analgesia is required (NRS score ≥4),iv fentanyl 25-50 mcg and/or ibuprofen and/or ketamine 10 mg will be administered. Patients are routinely administered iv dexamethasone 4 mg and IV 8 mg ondansetron 20 minutes before end of surgery for postoperative nausea and vomiting prophylaxis.
  Postoperative chronic pain will be assessed using the Brief Pain Inventory(BPI).
  Anxiety and depression status will be evaluated using the Hospital Anxiety and Depression Scale (HADS) .
  The character of pain will be evaluated using the Douleur Neuropathique 4 (DN4) score.
  Other Names: control
  Arms: Group Control
Drug: morphine PCA — V PCA of 0,5mg/ml morphine (the bolus dose is 20 µg/kg, the lock-in time of 6-10 minutes, the 4-hour limit is adjusted to be 80% of the calculated total amount).
  Other Names: PCA
  Arms: Group Control

SUMMARY:
The aim of this study is to investigate the effect of bilateral erector spinae plane (ESP) block application on postoperative chronic pain in patients undergoing on-pump open-heart surgery. At 3 months post-discharge, patients will be contacted by phone to assess their chronic pain status. Pain intensity and status will be evaluated using the Brief Pain Inventory, and the character of pain will be assessed using the Douleur Neuropathique 4 (DN4) score. Additionally, the patient's anxiety and depression status will be evaluated using the Hospital Anxiety and Depression Scale.

DETAILED DESCRIPTION:
Acute or chronic pain following cardiac surgery is a common issue that significantly impacts quality of life. The reported incidence of moderate to severe acute pain post-cardiac surgery varies widely in the literature, ranging from less than 5% to over 80%. Factors contributing to severe postoperative pain after median sternotomy include vasospasm, increased inflammatory response, soft tissue and bone injury during dissection, and chest tube placement. While pain typically decreases after the first 24 hours post-surgery, inadequate pain management can prolong this period. Chronic pain syndrome following sternotomy has been reported in 7% to 66% of patients undergoing open-heart surgery.

Initially, neuraxial anesthesia techniques such as thoracic epidural or thoracic paravertebral blocks were recommended for postoperative pain control in minimally invasive cardiac surgery. However, debates exist due to technical and patient-related challenges such as procedural difficulties, coagulation disorders, complete heparinization, hemodynamic instability, and pneumothorax. Fascial plane chest wall blocks involving serratus anterior and erector spinae have gained popularity for managing postoperative pain after minimally invasive cardiac surgery and thoracotomy/sternotomy, especially in patients receiving antiplatelet and anticoagulant therapy. An alternative approach, ultrasound-guided erector spinae plane block (ESPB), was introduced by Forero and colleagues in 2016 for treating thoracic neuropathic pain.

Inadequate pain control post-surgery can lead to persistent postoperative pain, high opioid consumption, and opioid-related morbidity. Theoretically, in patients receiving an erector spinae plane (ESP) block, the local anesthetic spreads both cranio-caudally and anteriorly through the costotransverse foramina, blocking the ventral/dorsal branches of spinal nerves, dorsal root ganglion, and rami communicantes at multiple levels. In patients undergoing sternotomy for cardiac surgery, bilateral thoracic ESP catheters or a single injection technique have reduced opioid use and pain scores.

This study is planned as a prospective, randomized controlled, double-blind, parallel-group trial.

Patients will be divided into two groups:

ESP Group: General anesthesia + ESP Block + Patient-Controlled Analgesia (PCA) Group K: General anesthesia + PCA

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 undergoing elective on-pump open-heart surgery via median sternotomy.
* American Society of Anesthesiologists (ASA)classification II-III patients.
* Patients who can use PCA.
* Patients who will sign the informed consent form.

Exclusion Criteria:

* History of opioid use for more than four weeks
* Chronic pain syndromes
* Patients with a history of local anesthetic or opioid allergy, hypersensitivity
* Alcohol and drug addiction
* Conditions where regional anesthesia is contraindicated
* Failure in the dermatomal examination performed after the block
* Emergency surgeries and redo surgeries.
* Individuals with obstructive sleep apnea.
* Left ventricular ejection fraction less than 30%.
* Patients with severe psychiatric illnesses (such as psychosis, dementia) that limit cooperation with verbal numerical pain scales.
* Pregnant and breastfeeding patients.
* Hematological disorders.
* Significant impairment in the function of a major organ (e.g., severe hepatic or renal disease).
* Patients who cannot be extubated within the first 6 hours postoperatively.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Chronic pain status | Postoperative 3rd month
  After patients are discharged, they will be contacted by phone at 3 months. Pain intensity and status will be assessed using the BPI, and the character of pain will be evaluated using the DN4 score.

SECONDARY OUTCOMES:
Postoperative opioid consumption in the first 24 Hours | Postoperative day 1
  Morphine consumption in the first 24 hours will be measured. Patients will be able to request opioids via a PCA device when their NRS score ≥4
Postoperative pain scores | Postoperative day 1
  Pain at rest and while coughing will be assessed by numerical rating scale (NRS) scores at 0, 3, 6, 12, 18, and 24 hours after extubation. The NRS is an 11-point numeric scale that ranges from 0 to 10. The NRS is an 11-point scale consisting of integers from 0 to 10: 0 indicates "no pain" and 10 indicates "the worst pain ever possible." One day before the surgery, all patients will be informed about NRS and instructed on how to use a patient-controlled analgesia device.
The incidences of post-operative nausea and vomiting (PONV) | Postoperative day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18, and 24 hours after extubation. If a score of 3 or more ondansetron 4 mg IV will be administered and will repeat after 8 hours if required.The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once.
The number of patient requiring rescue analgesic | Postoperative day 1
  The number of patients who required rescue analgesics will be recorded at 0, 3, 6, 12, 18, and 24 hours after extubation
Time to extubation | Postoperative day 1
  After the operation, the time until the patient is extubated will be recorded.
The number of patients with complications | Postoperative 7 days on an average
  The number of patients have any complications -directly related to the block or the drug used in the block- will be recorded.
Chronic pain status at 6 months. | Postoperative 6th month
  After discharge, patients will be contacted by phone at 6 months. Pain intensity and status will be assessed using the Brief Pain Inventory, and the character of pain will be evaluated using the Douleur Neuropathique 4 (DN4) score. Additionally, the patient's anxiety and depression status will be assessed using the Hospital Anxiety and Depression Scale.
Length of stay in the ICU | The time from admission to the ICU to the time of discharge to the hospital ward; during the hospital stay, an average of 7 days
  Total duration of stay in ICU will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Burhan Dost, Study Director — : Ondokuz Mayis Universitesi, Samsun, Atakum 55139
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No